CLINICAL TRIAL: NCT07049042
Title: Hypogonadotrophic Hypogonadism in Genetic Neurodevelopmental Conditions
Status: Recruiting | Type: Observational
Sponsor: University of Sheffield (Other)
Responsible Party: Sponsor
Other Study IDs: 340777
Record Dates: First submitted 2024-02-15; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Genetic Neurodevelopmental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hypogonadism is the medical name for a condition in which levels of the hormones which control sexual development are lower than normal. There are dozens of different causes of hypogonadism. Many people with hypogonadism have a change in a gene. There are many genes that give instructions for the hormones important for sexual development. Changes in one of these genes that stops the gene from working, can cause hypogonadism. In some of these medical conditions, there are additional features such as learning problems. In this study we will search databases to find all the genetic conditions that can be associated with hypogonadism. We will ask a number of people with changes in certain genes, identified from our search, to come to our research clinic. We will ask them about their health and examine them for signs of hypogonadism. For some, we will take blood samples to test for hypogonadism. This project will help us understand how common hypogonadism is, in people with these genetic changes, which will help with their treatment.

ELIGIBILITY:
Inclusion Criteria:

Pathogenic SNV or CNV in neurodevelopmental disorders gene of interest parent or carer consents to study

Exclusion Criteria:

parent or carer does not consent to study

Ages: 0 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with pathogenic CNVs or SNVs in a gene causing a neurodevelopmental disorder.
  Especially SOX genes to investigate association with hypogonadism.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2029-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of FSH | within 1 month of recruitment
  Blood sample to measure FSH levels.
  FSH (IU/l) reference range Male, female 0 - 1 month <22.0 Roche 24.01.2011 Male 1 month - 6 years <2.8 Roche 24.01.2011 Male 6 - 11 years <3.8 Roche 24.01.2011 Male 11 - 14 years <4.6 Roche 24.01.2011 Male 14 years + 1.5 - 12 Roche 24.01.2011 Females 1 month - 14 years 0 - 11 Roche 24.01.2011 Follicular phase 3.5 - 13 Roche 24.01.2011 Mid-cycle 4.7 - 22 Roche 24.01.2011 Luteal phase 1.7 - 7.7 Roc
Measurement of LH | within 1 month of recruitmen
  Blood sample to assay LH levels. LH (IU/l) reference range Males 0 - 1 year <3.2 Wiedemann Males 1 - 11 years <1.4 Roche 24.01.2011 Males 11 - 14 years <7.8 Roche 24.01.2011 Males 14 - 17 years 1.3 - 9.8 Roche 24.01.2011 Males 17 years + 1.7 - 8.6 Roche 24.01.2011 Females 0 - 6 years <0.5 Roche 24.01.2011 Females 6 - 11 years <3.1 Roche 24.01.2011 Females 11 - 14 years <11.9 Roche 24.01.2011 Follicular Phase 2.4 - 13 Roche 24.01.2011 Mid - cycle 14 - 96 Roche 24.01.2011 Luteal phase 1.0 - 11 Roche 24.01.2011 Females 60y + (post-menopausal) 7.7 - 59 Roche 24.01.2011
Measurement of testosterone. | within 1 month of recruitment.
  Blood assay of testosterone levels in males. Testosterone (nmol/l) Reference range Males, 6 months - 6 years <1.12 Roche 24.01.2011 Males 6 - 13 years <2.37 Roche 24.01.2011 Males 13 - 18 years 0.98 - 38.5 Roche 24.01.2011 Males 18 - 50 years 8.6 - 29 Roche 24.01.2011 Males 50 years + 6.7 - 25.7 Roche 24.01.2011 Females 0 - 1 month 0.7 - 2.2 Soldin 24.01.2011 Females 1 month - 10 years <0.4 Soldin 24.01.2011 Females 10 - 12 years <0.9 Soldin 24.01.2011 Females 12 years + 0.3 - 1.7 Roche 24.01.2011 Females 50 years + 0.1 - 1.4 Roche 24.01.2011
Physical examination for pubertal staging. | within 1- month of recruitment.
  Tanner staging standard exam (testicular volume, body hair development, breast development).
General medical examination. | within 1 month of recruitment
  Height & weight, dysmorphology exam. Full respiratory, cardiac and neurological exam.
Bone age from x-ray. | within 1-month of recruitment.
  X-ray assessment of bone age retrieved from medical notes (optional, only if done in routine clinical care previously).
Brain MRI | within 1 month of recruitment
  Result retrieved from medical records, optional only if done as part of routine care.
Gonadal ultrasound | within 1-month of recruitment
  gonadal ultrasound, optional, if done by usual care team
Serum oestradiol | within 1 month of recruitment
  Oestradiol (pmol/l) reference range Males 1 - 10 years 18.4 - 73.4 Roche 24.01.2011 Males aged 10 years + 41.4 - 159 Roche 07/09/2017 Females aged 1 - 10 years 22 - 99.1 Roche 24.01.2011 Follicular phase <91.8 - 854 Roche 02/08/2016 Ovulation phase 151 - 1461 Roche 02/08/2016 Luteal phase <91.8 - 1251 Roche 02/08/2016 Females post-menopausal <386 STH study 02/08/2016
Serum AMH | within 1 month of recruitment
  AntiMullerian Hormone (pmol/l) 2.5th, 5th , Median, 95th
  , 97.5th 20 - 24 yr 8.7, 10.9, 28.6, 71.0, 83.6 Roche 01/06/2018 25 - 29 yr 6.4, 8.6, 23.6, 64.6, 70.3 Roche 01/06/2018 30 - 34 yr 4.1, 5.1, 20.0, 54.2, 58.0 Roche 01/06/2018 35 - 39 yr 1.1, 2.9, 14.2, 49.7, 53.5 Roche 01/06/2018 40 - 44 yr 0.419, 0.4, 6.3, 31.7, 39.1 Roche 01/06/2018 45 - 50 yr 0.07, 0.07, 1.39, 12.8, 19.3 Roche 01/06/2018
Serum thyroid function tests | within 1 month of recruitment
  Free T3 (pmol/l) reference ranges Males, females 0 - 6 days 2.7 - 9.7 Roche 24.01.2011 Males, females 6 days - 3 months 3.0 - 9.3 Roche 24.01.2011 Males, females 3 - 12 months 3.3 - 9.0 Roche 24.01.2011 Males, females 1 - 6 years 3.7 - 8.5 Roche 24.01.2011 Males, females 6 - 11 years 3.9 - 8.0 Roche 24.01.2011 Males, females 11 - 20 years 3.9 - 7.7 Roche 24.01.2011 Males, females 20 years + 3.1 - 6.8 Roche 24.01.2011 Pregnancy, first trimester 3.8 - 6.0 Roche 24.01.2011 Pregnancy, second trimester 3.2 - 5.5 Roche 24.01.2011 Pregnancy, third trimester 3.1 - 5.0 Roche 24.01.2011 Free T4 (pmol/l) Males, females 0 - 6 days 11.0 - 32.0 Roche 24.01.2011 Males, females 6 days - 3 months 11.5 - 28.3 Roche 24.01.2011 Males, females 3 - 12 months 11.9 - 25.6 Roche 24.01.2011 Males, females 1 year + 11.9 - 21.6 Roche 14.03.2023 Pregnancy, first trimester 12.1 - 19.6 Roche 24.01.2011 Pregnancy, second trimester 9.6 - 17 Roche 24.01.2011 Pregnancy, third trimester 8.4 - 15.6 Roche 24.01.2011
Serum IGF1 level | within 1 month recruitment
  GF-1 (µg/l) Males, 0 - 3 months No range (comment) 06.10.2020 Males, 3 - 6 months 12 - 94 Roche 06.10.2020 Males, 6 - 12 months 12 - 95 Roche 06.10.2020 Males, 1 year 12 - 96 Roche 06.10.2020 Males, 2 years 14 - 104 Roche 06.10.2020 Males, 3 years 19 - 116 Roche 06.10.2020 Males, 4 years 27 - 134 Roche 06.10.2020 Males, 5 years 37 - 156 Roche 06.10.2020 Males, 6 years 47 - 184 Roche 06.10.2020 Males, 7 years 58 - 216 Roche 06.10.2020 Males, 8 years 68 - 254 Roche 06.10.2020 Males, 9 years 77 - 296 Roche 06.10.2020 Males, 10 years 86 - 343 Roche 06.10.2020 Males, 11 years 94 - 392 Roche 06.10.2020 Males, 12 years 101 - 434 Roche 06.10.2020 Males, 13 years 108 - 467 Roche 06.10.2020 Males, 14 years 115 - 489 Roche 06.10.2020 Males, 15 years 120 - 501 Roche 06.10.2020 Males, 16 years 125 - 503 Roche 06.10.2020 Males, 17 years 129 - 495 Roche 06.10.2020 Males, 18 years 132 - 476 Roche 06.10.2020 Males, 19 years 134 - 450 Roche 06.10.2020 Males, 20 years 136 - 421 Roche 06.10.2020 Males, 2
Serum prolactin | within 1-month recruitment
  Males, females 0 - 1 year No range (comment) Males 1 year + 86 - 324 Roche 24.01.2011 Females 1 year + 102 - 496 Roche 24.01.2011
serum cortisol | within 1 month recruitment
  Cortisol (nmol/l) Neonates 50 - 300 Sippell et al 01.06.2012 Adults 6 - 10 am 4 - 8 pm
  Random or 8.30-9.30 am:
  Adrenal insufficiency unlikely (NB does not apply to sick patients with high index of suspicion)
  Synacthen test (30 min cort):
  Primary adrenal insufficiency unlikely 133 - 537 68 - 327
  >/=350 >430 Wythenshawe In-house In-house 18.04.2016 21/12/2018 21/12/2018
serum ACTH | within 1-month
  ACTH, 7 am - 10 am (ng/l) 7.2 - 63.3 Roche 22/10/2018

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Childrens Hospital NHS Foundation Trust, Sheffield, Select, United Kingdom

IPD SHARING:
Plan to Share IPD: No